CLINICAL TRIAL: NCT05822063
Title: The Effect of Cold Packs, Lidocaine and Flash Lights on Cannulation Pain in Hemodialysis
Brief Title: The Effect of Cold Packs, Lidocaine and Flash Lights on Cannulation Pain in Hemodialysis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Farid, lecturer in clinical pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FAMASU/2023
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Arteriovenous Graft Site Pain
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lidocaine group (Active Comparator): the skin site will be prepped first and then two puffs of lidocaine (20 mg) will be sprayed by the researcher from a 5-cm distance on the dermal surface near the needle insertion point. Five minutes after spraying, the skin surface at the site of arterial needle insertion will be disinfected with 70% alcohol-soaked cotton pads and the specific hemodialysis needles will be inserted into the vessels of the fistula area by the ward nurse
  Interventions: Drug: Lidocaine topical
- cold packs (Active Comparator): In the ice pack method, 5 pieces of ice measuring 5*5 will be placed in latex gloves and covered with material cover. They were placed after the passage of 2 min on the hand at the site of fistula 5 min before making the puncture. Next, specific hemodialysis needles will be inserted in the vessels of fistula area by the ward nurse after disinfecting the fistula area with 70% alcohol-soaked cotton pads.
  Interventions: Other: cold packs
- flash lights (Active Comparator): the patient's face will be photographed. The photograph will be taken with a camera [(Sony HVLHFL1 with luminance intensity approximately 100 cd, lighting distance approximately 11 Lux, flash shooting distance (1-5 m)].
  Interventions: Device: flash lights
- control (No Intervention): no intervention

INTERVENTIONS:
Drug: Lidocaine topical — lidocaine spray
  Other Names: lidocaine spray
  Arms: Lidocaine group
Other: cold packs — ice packs
  Arms: cold packs
Device: flash lights — flash lights by camera
  Arms: flash lights

SUMMARY:
Compare the effects of lidocaine ,ice packs and flash lights on the intensity of pain induced by arteriovenous cannulation in hemodialysis patients.

DETAILED DESCRIPTION:
Chronic dialysis requires access to safe vessels that can be used for months; therefore, an arteriovenous fistula [AVF] is an appropriate option. Despite positive points, AVF has some disadvantages in comparison with other vascular access methods, including the inevitable pain of needle insertion in the fistula Each dialysis patient undergoes dialysis of approximately 3 times a week and 3 to 4 hours each time, which inevitably tolerates the pain caused by AVF cannulation 3 times a week. This pain will accompany these patients until the end of life unless they perform kidney transplantation

Half of dialysis patients express dissatisfaction with the experience of various types of pain, especially pain caused by AVF cannulation Reports have shown that 47% of dialysis patients, in addition to fear of cannulation pain, expressed this stage as the most stressful part of dialysis The main cause of this fear and apprehension is the diameter and length of the needle used for cannulation Repeated pain induced by hemodialysis fistula cannulation may lead to depression, reduced quality of life, pain, discomfort, distress, and stress, while controlling the pain improves the patients' acceptance of hemodialysis and their quality of life Considering the significance of pain, algesia relief must be considered as one part of treatment in these patients Presently, there is no uniform method to be used for relieving arteriovenous fistula cannulation pain in patients undergoing hemodialysis (Nasirzadeh, MircheraghI et al. 2019). There are various pharmacologic and nonpharmacologic modalities for pain relief. The effectiveness of some of these methods in relieving pain is still in under question.

Some of the puncture-related pain relief methods reported in literature include the application of heat or cold, EMLA local anesthesia creams, distraction methods, lidocaine gel, and lavender aroma inhalation

Ice pack and EMLA cream are two examples of local anesthetics which are readily applicable by the patients themselves . Ice is cheap and easily available with rapid and simple use which decreases pain by attenuating the signals of pain sensation, increasing perception of cold sensation instead of pain, and reducing the speed of neural transmission with pain neural fibers Lidocaine is one of the important common agents used as a local anesthetic . Lidocaine spray is one of the common formulations used clinically with moderate-term effect to induce local anesthesia in mucous membranes and skin. Depending on the site of application, anesthesia is usually induced during 1-5 min lasting for 10-15 min The EMLA cream as a local anesthetic contains lidocaine 25 mg/g and prilocaine 25 mg/g with little complications like slight redness of the site. It produces anesthesia of 5 mm depth . The theory behind pain reduction by lidocaine is the blocking of active and inactive sodium channels resulting in blockade of conduction and absence of stimulation followed by impaired or reduced pain transmission

Cutaneous stimulation includes cryotherapy thermotherapy, massage, pressure, and vibration, may help patients to relax or distract them from their pain. The term cryotherapy comes from the Greek ward cryo means cold and therapy means cure. Cryotherapy is the application of superficial cold & it is considered as a best cutaneous stimulation technique in terms of pain reduction. Applying cold will numb the area providing pain relief, reduce swelling and decrease metabolic rate reducing the oxygen requirements of the injured cells In the recent literature, venous cannulation pain after a flash of light has been shown to reduce the pain. During pain conditions, thalamic stimulation causes modulation of nociceptive information, leading to a reduction in pain perception. Thalamus is an integral part of the light reflex; it was presumed that a flash of light, by initiating a light reflex, might cause thalamic stimulation and thus decrease venous cannulation pain

Considering the contradictory results of these studies and regarding the importance of pain control in hemodialysis patients, this study explored the effect of lidocaine-containing compounds , ice pack, flash lights on the intensity of pain induced by arteriovenous cannulation in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will be willing to participate in the study.
2. Patients who are diagnosed as chronic kidney disease & undergoing haemodialysis with A.V. fistula of upper extremity currently used for haemodialysis which can be radio cephalic, radio basilic or brachio cephalic.
3. Chronic kidney disease patients who are visiting regularly, minimum 2 times per week for haemodialysis.

Exclusion Criteria:

1. Chronic kidney disease patients who are undergoing haemodialysis with other vascular access than A.V. fistula access.

4. Patients who are allergic to cold therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2023-08-25 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) | one month ( 30 days)
  it is score 1 to 10 according to pain intensity( 1= better ,10= worst)

IPD SHARING:
Plan to Share IPD: No